CLINICAL TRIAL: NCT05683210
Title: Comparison of The Effects of Initial Oral Feeding by Cup and Bottle-Feeding on Physiological Characteristics and Feeding Performance of Preterm Intants
Brief Title: Comparison of The Effects of Initial Oral Feeding by Cup and Bottle-Feeding of Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sukran Musaoglu, Nurse, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: cup and bottle feeding
Record Dates: First submitted 2023-01-03; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Oxygen Saturation; Heart Rate; Nutritional Status
Keywords: preterm infants; oxygen saturation; heart rate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cup feeding (Experimental): The infants in the control group were fed with a cup. During feeding, all infants in this group were placed in semi-elevated supine position. The position of the infant was adjusted so that when the milk reached the tongue, the infant would start foraging, dip his/her tongue into the milk by dimpling and slurp the milk with his/her tongue through a negative pressure, swallow as much as he/she wants and leave the rest back to the cup. The stopwatch was activated when the infant began to drink the milk from the cup, and the stopwatch was stopped when the infant no longer slurped the milk, and the feeding process was completed. When the infant was physiologically (HR of 120-160/min, SpO2 ≥90) and behaviourally ready, feeding was resumed and the infant was prevented from getting tired during feeding and actively participated in feeding. Feeding time was limited to 30 minutes in either group, including the infants' resting time.
  Interventions: Behavioral: Cup feeding
- Bottle feeding (Experimental): The infants in the experimental group were fed with a bottle. The teat of the feeding bottle was selected to be smaller in size, softer and with a smaller hole than the teat of the term infant and suitable for preterm infants. The same brand and model of bottle and teat were used for each infant. All infants in this group were fed in a semi-elevated side-lying position, as it was more similar to the position in which the infant suckled the mother's breast. The infant's lips were tapped with the bottle teat for stimulating to feed, and when the infant opened his/her mouth and drooped his/her tongue, the teat of the bottle was put into his/her mouth. The time elapsed from when the infant started to suck the bottle until he/she released the bottle from his/her mouth was considered as the feeding phase.
  Interventions: Behavioral: Bottle feeding

INTERVENTIONS:
Behavioral: Cup feeding — The preterm infant was put on pulse oximetry and monitored, and heart rate and oxygen saturation began to be monitored. The infants' heart rate and oxygen saturation were recorded 30 minutes before feeding, and their signs of preparedness for oral feeding were monitored. After the data were recorded for 30 minutes, the infant was taken out of the incubator and his/her body weight was measured naked with only a clean diaper to determine the test weight. Feeding time was limited to 30 minutes, including the infants' resting time. When the infant was no longer sucking, the stopwatch was stopped, and the feeding phase was terminated. The feeding process was completed at the end of 30 minutes even if the infant did not take all of the food. The infant was followed up for 30 minutes after the end of feeding. During this time, the pulse oximetry continued to record and no intervention was made in order to avoid any effect on physiological values.
  Arms: Cup feeding
Behavioral: Bottle feeding — The preterm infant was put on pulse oximetry and monitored, and heart rate and oxygen saturation began to be monitored. The infants' heart rate and oxygen saturation were recorded 30 minutes before feeding, and their signs of preparedness for oral feeding were monitored. After the data were recorded for 30 minutes, the infant was taken out of the incubator and his/her body weight was measured naked with only a clean diaper to determine the test weight. During the feeding period, heart rate and oxygen saturation were continuously recorded. Feeding time was limited to 30 minutes, including the infants' resting time. When the infant was no longer sucking, the stopwatch was stopped, and the feeding phase was terminated. The infant was followed up for 30 minutes after the end of the feeding. During this time, the pulse oximetry continued to record and no intervention was made in order to avoid any effect on physiological values.
  Arms: Bottle feeding

SUMMARY:
The research was planned in a randomized controlled experimental design to determine the effects of the cup and bottle used during the first oral feeding on physiological characteristics and feeding performance in preterm infants. The research was carried out between January 2021 and February 2022 at the Neonatal Intensive Care Unit of Göztepe Süleyman Yalçın City Hospital. Research data were obtained from preterm infants who were born before 34 weeks of gestation, appropriate to selection of study group criterias and hospitalized in the neonatal intensive care unit. A total of 80 babies in the sample group were randomly assigned to the experimental (bottle) and control (cup) groups. Oxygen saturation, heart rate, feeding performance and test weight before, during and after feeding of preterms in both groups were compared. There was no statistically significantly difference between the experimental and control groups in terms of oxygen saturation and heart rate.

DETAILED DESCRIPTION:
The coordination of sucking, swallowing and breathing is necessary for the preterm infant to be effectively and safely fed by the oral route. Although the sucking motion begins in the 27-28th week, the coordination of sucking, swallowing, and breathing appears in the 32-34th week. Introducing oral feeding to preterm infants is recommended by sucking the mother's breast when they are ready for oral feeding. Preterm infants are fed through complementary feeding methods such as a bottle, spoon, dropper, cup, and finger feeding until they reach the condition to meet their nutritional needs by sucking the mother's breast.

Bottle feeding is one of the nutritive sucking methods commonly used in both preterm and term infants worldwide. When the mother is unable to breastfeed or breast milk is not available, preterm infants can be fed with a bottle. Bottle feeding contributes to effective feeding and helps the infant to relax by meeting the sucking reflex. Cup feeding has been used in developed and developing countries for many years to feed premature infants and those with low birth weights. Cup feeding is a simple, practical, effective, and low cost method that can be used in infants who can swallow but are unable to suck well enough to be fed completely from the mother's breast, and in cases where an alternative such as a gastric catheter or a bottle is required for feeding.

Studies that compared bottle and cup feeding reported that the swallowing performance of preterm infants fed with a bottle was better, the length of hospital stay was longer in preterm infants fed with a cup, and the duration of feeding was longer in preterms fed with a cup compared to those fed with a bottle, the rate of breastfeeding after discharge was higher in those fed with a cup, no significant difference was found in weight gain, but the quantity of food intake was less and the rate of food spillage was higher in preterm infants fed with a cup compared to those fed with a bottle. For all of these reasons, bottle feeding is reported to be a safer and more appropriate method.

This randomised controlled experimental study was carried out to compare the effect of cup and bottle feeding on physiological characteristics and feeding performance in preterm infants born at or below the 34th gestational week. A power analysis was used to determine. The study included a total of 80 preterms, 40 preterms for each group. The parents of preterm infants who met the inclusion criteria granted their written and verbal consent.

Experimental Group

The preterm infant was put on pulse oximetry and monitored, and heart rate and oxygen saturation began to be monitored. No invasive intervention or care was provided for the infant to rest for 1 hour before feeding. Data were collected during working hours (08.00-16.00) to establish common physical environment conditions for each infant. Bottles and teats to be used during feeding were sterilised with a steam steriliser. The heart rate and oxygen saturation of the infants were recorded 30 minutes before the time of feeding, and their signs of preparedness for oral feeding were monitored. After the data were recorded for 30 minutes, the infant was taken out of the incubator and his/her body weight was measured naked with only a clean diaper to determine the test weight. All findings were recorded on the "Feeding Monitoring Form".

After all steps before feeding were completed and recorded, the infant was loosely wrapped with a soft cloth and started to be fed by being held only by the researcher in order to prevent the effect of different feeding practices of the nurses on the study. As soon as feeding was initiated, a stopwatch was activated by another nurse who worked in the clinic in order to avoid any bias, and the feeding time was maintained not to exceed 30 minutes to prevent the infant from getting tired. During the feeding period, heart rate and oxygen saturation were continuously recorded. The infants in the experimental group were fed with a bottle. The teat of the feeding bottle was selected to be smaller in size, softer and with a smaller hole than the teat of the term infant and suitable for preterm infants. The same brand and model of bottle and its teat were used for each infant. All infants in this group were fed in a semi-elevated side-lying position, as it was more similar to the position in which the infant suckled the mother's breast. The infant's lips were tapped with the bottle teat for stimulating to feed, and when the infant opened his/her mouth and drooped his/her tongue, the teat of the bottle was put into his/her mouth. During feeding, stimulant behaviours such as pushing the bottle back and forth and swirling the bottle in the mouth were avoided in order to allow the infant to suck faster and accelerate the flow. The time elapsed from when the infant started to suck the bottle until he/she released the bottle from his/her mouth was considered as the feeding phase.

Physiological and behavioural signs of stress (throwing the head backwards, trying to push the bottle and cup away with the tongue, arching back, grimacing, fanning the fingers, rapid and loud breathing, aspiration, coughing and trying to swallow quickly, desaturation (<90), apnoea, tachycardia, bradycardia and colour change) were observed in all bottle and cup-fed infants during feeding. Also, signs of fatigue (i.e., decreased muscle tone, inability to maintain flexion posture, reduced sucking-swallowing activity, spilling milk out of the mouth) were observed in both groups.

In case of signs of stress and fatigue, feeding was interrupted for a short time and the infant was allowed to rest. When the infant was physiologically (HR of 120-160/min, SpO2 ≥90) and behaviourally ready, feeding was resumed and the infant was prevented from getting tired during feeding and actively participated in feeding. Feeding time was limited to 30 minutes, including the infants' resting times. When the infant was no longer sucking, another nurse who worked in the clinic stopped the stopwatch in order to prevent bias and the feeding phase was terminated. The feeding process was completed at the end of 30 minutes even if the infant did not take all of the food.

After feeding, the body weight of the infants was measured only with the diaper on and the test weight was determined. Test weighing is a technique used to measure the amount of nutrition of the infant, in which the infant is weighed before and after feeding without undressing if the infant is dressed and without changing the diaper if the infant is diapered, and 1 gram corresponds to 1 ml of breast milk. After the procedure, the infant was put in the incubator in a right-side position to facilitate gastric discharge. The infant was followed up for 30 minutes after the end of the feeding. During this time, the pulse oximetry continued to record and no intervention was made in order to avoid any effect on physiological values. The recorded data were classified into pre-feeding, feeding and post-feeding periods, entered into a computer environment, and averaged. The amount of food taken by the infant during the 30-minute feeding was recorded, and if the infant was unable to take the entire amount of food prescribed by the physician, he/she took the remaining amount with an orogastric catheter after the post-feeding measurements were finished.

Control Group

The preterm infant was put on pulse oximetry and monitored, and heart rate and oxygen saturation began to be monitored. No invasive intervention or care was provided for the infant to rest for 1 hour before feeding. Data were collected during working hours (08.00-16.00) to establish common physical environment conditions for each infant. The cup to be used during feeding was sterilised with a steam steriliser. The heart rate and oxygen saturation of the infants in both groups were recorded 30 minutes before the time of feeding and their signs of preparedness for oral feeding were monitored. After the data were recorded for 30 minutes, the infant was taken out of the incubator and his/her body weight was measured naked with only a clean diaper to determine the test weight. All findings were recorded on the "Feeding Monitoring Form".

After all steps before feeding were completed and recorded, the infant was loosely swaddled with a soft cloth and started to be fed by being held only by the researcher in order to prevent the effect of different feeding practices of the nurses on the study. As soon as feeding was initiated, a stopwatch was activated by another nurse who worked in the clinic in order to avoid any bias, and the feeding time was maintained not to exceed 30 minutes in order to prevent the infant from getting tired. During the feeding period, heart rate and oxygen saturation were continuously recorded. The infants in the control group were fed with a cup. The cups currently used in the clinic for feeding were selected in a size suitable for the preterm infant so that they would not damage the lips, palate and tongue. During feeding, all infants in this group were placed in semi-elevated supine position. The cup was inserted into the infant's lips and elevated until the milk reached the infant's mouth. The position of the infant was adjusted so that when the milk reached the tongue, the infant would start foraging, dip his/her tongue into the milk by dimpling and slurp the milk with his/her tongue through a negative pressure, swallow as much as he/she wants and leave the rest back to the cup. The cup was not raised to allow the infant to slurp the milk more quickly and the milk was not poured into his/her mouth, so that the infant was given complete control over the feeding. The stopwatch was activated when the infant began to drink the milk from the cup, and the stopwatch was stopped when the infant no longer slurped the milk, and the feeding process was completed. In case of signs of stress and fatigue, feeding was interrupted for a short time and the infant was allowed to rest. When the infant was physiologically (HR of 120-160/min, SpO2 ≥90) and behaviourally ready, feeding was resumed and the infant was prevented from getting tired during feeding and actively participated in feeding. Feeding time was limited to 30 minutes, including the infants' resting times. When the infant was no longer sucking, another nurse who worked in the clinic stopped the stopwatch in order to prevent bias and the feeding phase was terminated. The feeding process was completed at the end of 30 minutes even if the infant did not take all of the food. After feeding, the body weight of the infants was measured with only the diaper on and the test weight was determined. After the procedure, the infant was put in the incubator in a right-side position to facilitate gastric discharge. The infant was followed up for 30 minutes after the end of feeding. During this time, the pulse oximetry continued to record and no intervention was made in order to avoid any effect on physiological values. The recorded data were classified into pre-feeding, feeding, and post-feeding periods, entered into a computer environment, and averaged. The amount of food taken by the infant during the 30-minute feeding period was recorded, and if the infant was unable to take in the entire amount of food prescribed by the physician, he/she took the remaining amount with an orogastric catheter after the post-feeding measurements were finished.

ELIGIBILITY:
Criteria for Sample Selection

* Being at the ≤34th gestational week according to the last menstrual period of the mother of the preterm
* Being at the ≥30th postmenstrual week on the date of inclusion in the study
* Having a body weight of 1000 grams or more on the date of inclusion in the study
* Switching from enteral feeding to oral feeding for the first time with the joint decision of the physician and nurse
* Breastfeeding
* Showing physiological and behavioural signs indicating that the infant is ready for oral feeding (tolerating full enteral feeding, exhibiting sucking behaviour, opening the mouth by responding to stimuli around the mouth, normal physiological values [HR of 120-160/min, SpO2≥90], maintaining alertness, keeping the body in flexion posture)
* Having parental consent for inclusion in the study and an informed consent form signed by parents

Exclusion Criteria

* Having diagnostic criteria for severe bronchopulmonary dysplasia (≥30% O2 requirement and/or positive pressure requirement at the 36th postmenstrual week or at discharge in preterm infants with a gestational age of <32 weeks; ≥30% O2 requirement or positive pressure requirement at the 56th postnatal day or at discharge in preterm infants with a gestational age of ≥32 weeks)
* Having an anomaly such as cleft palate, cleft lip
* Having gastrointestinal, neurological or genetic disease (NEC, IVH, hydrocephalus, asphyxia, Down syndrome, short bowel syndrome, etc.)

Ages: 30 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Feeding Status | maximum 30 minutes
  In order to assess the feeding status of the infant, his/her time of feeding and the amount of nutrient he/she receives in a minute will be calculated. In order to determine his/her time of feeding, a phone chronometer will be started as soon as he/she begins feeding and it will be stopped when feeding is over. All infants in experimantal group and control group will be fed with a slow-flow bottle branded Avent which is designed for premature infants. It will be calculated how much (cc) of the total amount of nutrient ordered by the doctor the infant receives. The total amount of nutrient received by the infant will be divided into the time of feeding and thus the amount of nutrient received in a minute (cc) will be calculated.

SECONDARY OUTCOMES:
Heart Rate | All babies in experimental group and control group will be recorded in the registration form by the observing nurse once half an hour before the feeding time, 30 minutes before the feeding time, during the feeding and at 30 minutes after the feeding.
  The "Covidien Nellcor Pulse Oximeter Bedside" device and its probe were employed to determine the heart rate of preterm infants before, during, and after feeding. Alert limits for heart rate were set as 120-160/min on the device. The heart rate of preterm infants in the experimental and control groups began to be recorded 30 minutes before feeding and continued to be recorded during the feeding and for 30 minutes after the end of the feeding.
Oxygen Saturation | All babies in experimental group and control group will be recorded in the registration form by the observing nurse once half an hour before the feeding time, 30 minutes before the feeding time, during the feeding and at 30 minutes after the feeding.
  The "Covidien Nellcor Pulse Oximeter Bedside" device and its probe were employed to determine oxygen saturation in preterm infants before, during and after feeding. The oxygen saturation below 90% for more than one second was considered as desaturation in the study. The oxygen saturation of preterm infants in the experimental and control groups began to be recorded 30 minutes before feeding and continued to be recorded during the feeding and for 30 minutes after the end of the feeding.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Gözen, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University, Cerrahpaşa, Istanbul, Turkey (Türkiye)